CLINICAL TRIAL: NCT02314767
Title: A Finnish Community Randomized Psychotherapy Effectiveness Study for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, HSaloheimo, MD Psychiatrist, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lohja Depression Treatment
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Interpersonal Psychotherapy (Active Comparator): Interpersonal Psychotherapy treatment for MDD patients was implemented with antidepressant pharmacotherapy by national Quidelines for the treatment of Patients with depression. Intervention:Interpersonal psychotherapy as ADD-on method. Outcome was compared with patients in treatment as usual group.
  Interventions: Behavioral: Interpersonal Psychotherapy; Behavioral: Psychoeducational Group Therapy
- Psychoeducational Group Therapy (Active Comparator): Psychoeducational Group Therapy arm for MDD patients with antidepressant pharmacotherapy by national Quidelines for the treatment of Patients with depression. Intervention: Psychoeducational Group Treatment as ADD-on method.
  Interventions: Behavioral: Interpersonal Psychotherapy; Behavioral: Psychoeducational Group Therapy
- Treatment as Usual (No Intervention): Treatment as usual ( consisting of supportive psychodynamic-oriented treatment) with antidepressant pharmacotherapy by national Quidelines for the treatment of Patients with depression

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Patients were treated with IPT method, which was an active comparator vs treatment as usual
  Arms: Interpersonal Psychotherapy; Psychoeducational Group Therapy
Behavioral: Psychoeducational Group Therapy — Patients were treated with PeGt method which was an active comparatos vs treatment as usual
  Arms: Interpersonal Psychotherapy; Psychoeducational Group Therapy

SUMMARY:
Lohja Depression Treatment Study is a randomized treatment trial which compares three approaches for treatment of depression:1) Interpersonal Psychotherapy (IPT), 2) Psychoeducational Group Treatment ( PeGT) and 3) Treatment as Usual (TAU). This Trial aims to test and adapt known short term treatment models for Finnish patients and circumstances.

DETAILED DESCRIPTION:
Patients having signs of depression referred to Lohja area secondary level psychiatric clinics were assessed to the trial. After verification the diagnosis of Major Depressive Disorder (MDD) they were informed of the study. Consented patients were randomized to three study arms.

Baseline clinical demographics was collected. Psychotherapeutic treatment was implemented by specially trained therapists and the study data was collected by trained psychiatrists who were blinded to the therapy model patients has received.Primary outcome measure was 17-item Hamilton Depression Rating Scale (HAMD) and secondary outcome measures were Clinical Global Impression scale (CGI), Social and Occupational Functioning Assessment Scale ( SOFAS), Social Adaptation Scale ( Finnish translation JES) and Quality of Life assessment ( a Finnish validated questionnaire 15-D).The total of sick leave days and number of possible disability pensions in a year were assessed as well.

Assessments were implemented at the beginning, at 1,5 month, at 3 months ( which was the end of active treatment of short-term psychotherapies), at 6 months and at 12 months.

The primary assessment was planned to carry out using tests of group comparison. Sample size of 32 and 32 achieve 91% power to detect a clinically meaningful difference with a significance level (alpha) of 0.01 using two-sided two-sample t-test. Baseline differences in demographic variables and the depression measurement across the three treatment groups were tested using chi-square tests and analysis of variance.Likelihood-based inference using linear mixed models were employed to analyze treatment effects, focusing on the time x treatment interaction. Separate analyses assessed IPT-TAU and PeGT-TAU comparisons. All statistical analyses were performed using R. The aim of this study was to get a total of 140-160 patients, about 50 patients on one group.The final number of patients showed to be 134.

The statistical calculation was intent-to-treat model with consideration to missing data, because in this kind of natural setting notable attrition was assumed. The training of the therapists and researchers and quality control during assessments was considered and personnel was supervised throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder - diagnosed
* Comorbid anxiety disorders

Exclusion Criteria:

* Psychosis
* Suicidal patients
* Serious acute somatic illness
* Inability to read and write
* alcohol dependence or use of illicit drugs

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2004-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hamilton Rating Scale for Depression at 12 months | 12 months

SECONDARY OUTCOMES:
Change from baseline Clinical Global Impression, severity and change at 12 months | 12 months
Change from baseline Social and Occupational Functioning Assessment Scale at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heikki O Katila, MD Ph.D., Study Director — University of Helsinki

REFERENCES:
- [Derived] Saloheimo HP, Markowitz J, Saloheimo TH, Laitinen JJ, Sundell J, Huttunen MO, A Aro T, Mikkonen TN, O Katila H. Psychotherapy effectiveness for major depression: a randomized trial in a Finnish community. BMC Psychiatry. 2016 May 6;16:131. doi: 10.1186/s12888-016-0838-1. PMID 27153942